CLINICAL TRIAL: NCT02026141
Title: Can Dexmedetomidine For Procedural Sedation In Knee Arthroplasty Reduce Postoperative Pain? A Randomized Control Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Ian Chan, MD, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UofS 13-232
Record Dates: First submitted 2013-12-29; First posted 2014-01-01 (Estimated); Results first posted 2016-06-20 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-05

CONDITIONS: Total Knee Arthroplasty
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexmedetomidine arm (Experimental): Standardized pre-op meds and spinal anesthetic.
  Once the patient's spinal is performed, patient will receive the following:
  Start with bolus of 0.5micrgram/kg over 10 minutes, and then infusion of 0.5 microgram/kg/hr
  Infusion will be stopped after the last staple or suture is performed on the incision.
  Both groups will have a midazolam 0.5mg prn q 5minutes to be used as a rescue to achieve moderate sedation as defined by ASA.
  Interventions: Drug: Dexmedetomidine
- Saline Placebo (Placebo Comparator): Patients will receive the standardized pre-op meds and spinal anesthetic. Once the spinal anesthetic is performed,
  Patient will receive the same infusion rates as in the Dexmedetomidine arm, however with Normal Saline as a Placebo.
  midazolam 0.5mg prn q 5minutes to be used as a rescue to achieve moderate sedation.
  Interventions: Drug: Normal Saline Placebo

INTERVENTIONS:
Drug: Dexmedetomidine
  Arms: Dexmedetomidine arm
Drug: Normal Saline Placebo
  Arms: Saline Placebo

SUMMARY:
Dexmedetomidine has been often used for procedural sedation. It has also has been shown to have a pain sparing effect. Therefore the investigators propose that if Dexmedetomidine is used for sedation in total knee replacements done under spinal anesthetic, the patients will have less pain up to 24 hours after the procedure.

DETAILED DESCRIPTION:
Randomization will occur prior to patient being brought into operating room (by pharmacy or by the anesthesia research coordinator). A third anesthetist not involved in the project will mix up the syringe based on instructions in an opaque envelope, and provide the syringe to the attending anesthetist.

The current standard of care entails patients receiving a midazolam bolus for sedation during the operation. The investigators propose to substitute a syringe of dexmedetomidine or saline to be run as an infusion throughout the case for sedation. A midazolam bolus will be available at anesthetist discretion to achieve a moderate sedation score as defined by the American Society of Anesthesia.

Standardized Medication Protocol

Pre-op:

Tylenol and Naproxen

Spinal:

Marcaine .75%, 1.7cc (12.75mg) Fentanyl 10 micrograms

Sedation

1. st arm- Dexmedetomidine, drawn up into a 50cc syringe of saline, thereby making it 5ug/ml.
2. nd arm- Receives Normal Saline syringe

Plan for bolus of 0.5microgram/kg over 10 minutes, and then infusion of 0.5 microgram/kg/hr (Can be titrated from 0.2-0.7 microgram per kg per hr to achieve moderate sedation as defined by the ASA

Both groups will have a midazolam 0.5mg prn q 5minutes to be used as a rescue to achieve moderate sedation.

Post op- Initial setting of patient-controlled-analgesia pump to be set at morphine 1 mg, lockout of 8 minutes, to be increased to 1.5 mg with lockout of 6 minutes if pain not controlled. The investigators will increase the pump dose by 0.5 mg/dose/1 hr until pain controlled.

Risks The most common treatment-emergent adverse reactions for dexmedetomidine, occurring in 2% of patients in both ICU and procedural sedation studies, include- Hypotension, Bradycardia and Dry mouth. To minimize the risks to participants, an anesthesiologist will always be present in the room while the infusion is running, will monitor the patient, and will be allowed to treat as they see fit any of these risks.

Data Collection Data collection will be performed primarily by Ian Chan, anesthesiology resident.

Primary Outcome:

Total morphine consumption in the first 24 hours

ELIGIBILITY:
Inclusion Criteria:

* Total Knee arthroplasty American Society of Anesthesiologist score of 1-3 Age 18-85 Elective total knee arthroplasty under spinal anesthetic.

Exclusion Criteria:

* Contraindication to Dexmedetomidine. (second or third degree heart block, renal or hepatic dysfunction) Contraindication to Spinal Anesthetic Pain being treated by opioids prior to operation Contraindication to premedication Previous total knee arthroplasty

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian A Chan, MD, Principal Investigator — Department of Anesthesia, University of Saskatchewan, Canada; Jurgen Maslany, MD, FRCPC, Principal Investigator — University of Saskatchewan; Kyle Gorman, MD, FRCPC, Principal Investigator — University of Saskatchewan
Locations (1):
- Regina General Hospital, Regina, Saskatchewan, Canada

REFERENCES:
- [Derived] Chan IA, Maslany JG, Gorman KJ, O'Brien JM, McKay WP. Dexmedetomidine during total knee arthroplasty performed under spinal anesthesia decreases opioid use: a randomized-controlled trial. Can J Anaesth. 2016 May;63(5):569-76. doi: 10.1007/s12630-016-0597-y. Epub 2016 Jan 29. PMID 26830642

RESULTS

PARTICIPANT FLOW:
Groups:
- Dexmedetomidine Arm: Standardized pre-op meds and spinal anesthetic.
  Once the patient's spinal is performed, patient will receive the following:
  Start with bolus of 0.5micrgram/kg over 10 minutes, and then infusion of 0.5 microgram/kg/hr Infusion will be stopped after the last staple or suture is performed on the incision.
  Both groups will have a midazolam 0.5mg prn q 5minutes to be used as a rescue to achieve moderate sedation.
  Dexmedetomidine
- Saline Placebo: Patients will receive the standardized pre-op meds and spinal anesthetic. Once the spinal anesthetic is performed,
  Patient will receive the same infusion rates as in the Dexmedetomidine arm, however with Normal Saline as a Placebo.
  midazolam 0.5mg prn q 5minutes to be used as a rescue to achieve moderate sedation.
  Normal Saline Placebo
Period: Overall Study
Arm/Group | Dexmedetomidine Arm | Saline Placebo
Started | 20 | 20
Completed | 20 | 19
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Dexmedetomidine Arm: Standardized pre-op meds and spinal anesthetic.
  Once the patient's spinal is performed, patient will receive the following:
  Start with bolus of 0.5micrgram/kg over 10 minutes, and then infusion of 0.5 microgram/kg/hr
  Infusion will be stopped after the last staple or suture is performed on the incision.
  Both groups will have a midazolam 0.5mg prn q 5minutes to be used as a rescue to achieve moderate sedation as defined by ASA.
  Dexmedetomidine
- Total: Total of all reporting groups
Arm/Group | Dexmedetomidine Arm | Saline Placebo | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 11 | 20
  >=65 years | 11 | 9 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (11.4) | 66.1 (8.2) | 66.2 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 12 | 28
  Male | 4 | 8 | 12
Region of Enrollment [Number; unit: participants]
  Canada | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Morphine Consumption
Description: Patients will be provided with a patient-controlled-analgesia in which they will have morphine available for pain scores greater than 3.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Dexmedetomidine Arm | Saline Placebo
Number analyzed (Participants) | 20 | 20
milligrams | 29.2 (11.2) | 61.2 (17.2)
Statistical Analysis 1: Comparison: Dexmedetomidine Arm vs Saline Placebo; Test type: Superiority or Other; p < 0.05, ANCOVA

2. Secondary Outcome: Time of First Analgesia Request
Time Frame: time of first analgesia request from closure of skin up to 24 hours.
Reporting Status: Not Posted

3. Other Pre Specified Outcome: VAS Scores
Description: Patients will be asked to chart their VAS pain score at the 6, 12 , and 24 hour mark.
Time Frame: 6, 12 and 24 hour marks.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Dexmedetomidine Arm | Saline Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No